CLINICAL TRIAL: NCT00187486
Title: Phase II Study of Tarceva Plus Temodar During and Following Radiation Therapy in Patients With Newly Diagnosed Glioblastoma Multiforme and Gliosarcoma
Brief Title: Safety and Efficacy Study of Tarceva, Temodar, and Radiation Therapy in Patients With Newly Diagnosed Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC 04101; OSI 2725s (Other: Genentech, Inc)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Glioblastoma Multiforme; Gliosarcoma
Keywords: Glioblastoma Multiforme; Gliosarcoma; GBM; GS; Tarceva; Temodar; Radiation; Newly Diagnosed
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Erlotinib Hydrochloride; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temodar plus Tarceva plus Radiation Therapy (Experimental): Single arm phase-2 experimental treatment of newly diagnosed patients with Glioblastoma with Temodar plus Tarceva plus Radiation Therapy
  Interventions: Drug: Tarceva; Drug: Temodar; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: Tarceva — Tarceva (erlotinib hydrochloride; previously referred to as OSI-774), a quinazoline, is an orally active, potent, selective inhibitor of EGFR tyrosine kinase. 100 - 300 milligrams (mg) every day (QD) orally (PO) every (q) 28 days depending on EIAED Status
  Other Names: erlotinib
Drug: Temodar — Temodar 200 mg/m^2/day x 5 days every 28 days
  Other Names: temozolomide
Procedure: Radiation Therapy — Radiotherapy will be administered in 180 centigray(cGy)/day - 200cGy/day fractions delivered 5 days per week to a total dose of 5940cGy - 6100cGy. A total of 4500cGy will be delivered to the clinical tumor volume consisting of T2-bright edema + a 2centimeter margin, or, if no edema, the contrast enhancing lesion +2.5 centimeter margin. An additional boost of 1440cGy will be delivered to the gross tumor volume consisting of the contrast enhancing lesion + a 1 centimeter margin.

SUMMARY:
The patients eligible for this study are those diagnosed with glioblastoma or gliosarcoma who have recently undergone surgery and who have not been treated with radiation therapy or chemotherapy. This is called a phase II study. The purpose of the phase II study is to determine how effective Tarceva plus Temodar plus radiation is in controlling the growth of glioblastoma and gliosarcoma. All patients will receive radiation and Temodar plus Tarceva. There is no "placebo" drug.

DETAILED DESCRIPTION:
This is a Phase II Study of Tarceva plus Temodar during and following radiation therapy in patients with newly diagnosed glioblastoma multiforme and gliosarcoma. The efficacy and safety profile of Tarceva in combination with radiation therapy plus Temodar will be studied. In addition, correlations between response to treatment and epidermal growth factor receptor (EGFR) status as well as other molecular markers of tumor prior to treatment will be explored. Patients will be stratified according to enzyme inducing anti epileptic drug (EIAED) use. Group A (not on EIAEDs) will take 100 milligrams (mg) Tarceva/day during radiotherapy and start with a dose of 150 mg Tarceva/day two weeks after radiotherapy. Group B (on EIAEDs) will take 200mg Tarceva/day during radiotherapy and start with a dose of 300 mg Tarceva/day two weeks after radiotherapy. Both groups will take 75 mg/m^2 Temodar/day during radiotherapy and 200 mg/m^2 Temodar/day x 5 two weeks after radiotherapy. Intrapatient Tarceva dose escalation may occur every two weeks after radiotherapy until the appearance of a particular rash severity. The maximum dose allowed is 200 mg for group A and 500 mg for group B.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven intracranial glioblastoma multiforme (GBM) and gliosarcoma (GS) will be eligible for this protocol.
* Diagnosis will have been established by biopsy or resection no more than 5 weeks prior to treatment.
* An magnetic resonance imaging (MRI) or computer tomography (CT) must be obtained within 14 days of treatment. The use of MRI rather than CT is preferred. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for assessment of tumor status.
* Patients without measurable or assessable disease are eligible.
* Patient must not have had prior cranial radiation therapy.
* Patients must not have received prior cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy for brain tumors.
* Patients who received Gliadel wafers at the time of original resection will be excluded.
* Patients must have a plan to begin partial brain radiotherapy the same day as Tarceva and temozolomide.
* Radiotherapy must be a) at the Radiation Oncology Department of the University of California San Francisco or b) at an affiliated site such that a radiation oncologist at UCSF can provide assurance that radiation can be performed as specified.
* Radiotherapy must be given by external beam to a partial brain field in daily fractions of 1.8 to 2.0 Gy, to a planned total dose to the tumor of 5940-6100 cGy.
* Stereotactic radiosurgery and brachytherapy will not be allowed.
* Patients must be willing to forego other cytotoxic and non-cytotoxic drug therapy against the tumor while being treated with Tarceva and temozolomide.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Patients must be registered in the UCSF Neuro-Oncology database prior to treatment with study drug.
* Patients must sign an authorization for the release of their protected health information.
* Patients must be 18 years or older, and with a life expectancy > 12 weeks.
* Patients must have a Karnofsky performance status of > 60.
* Patients must have adequate bone marrow function (WBC > 3,000/µl, ANC > 1,500/mm^3, platelet count of > 100,000/mm^3, and hemoglobin > 10 gm/dl), adequate liver function (SGOT, and bilirubin < 2 times ULN), and adequate renal function (creatinine < 1.5 mg/dL or calculated creatinine clearance > 60 cc/min) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race.
* Patients must not have active infection.
* Patients must not be pregnant/breast feeding and must agree to practice adequate contraception.
* Women of childbearing potential must have a negative B-HCG pregnancy test documented within 7 days prior to registration.
* Patients must not be pregnant because of the uncertainty that study drug may be potentially embryotoxic. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation, and continue approximately 12 weeks after the study is completed. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.
* Patients must not have serious inter-current medical illness.
* Patient with recent thromboembolic disease (deep vein thrombosis and pulmonary embolism) are eligible if they are clinically stable and the thromboembolic event occurred more than 3 weeks prior to enrollment into this protocol.

Exclusion Criteria:

* Patients who do not meet one or more of the inclusion criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2004-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Prados, MD, Principal Investigator — UCSF Department of Neurological Surgery
Locations (1):
- UCSF Department of Neurological Surgery, San Francisco, California, United States

REFERENCES:
- [Result] Prados MD, Chang SM, Butowski N, DeBoer R, Parvataneni R, Carliner H, Kabuubi P, Ayers-Ringler J, Rabbitt J, Page M, Fedoroff A, Sneed PK, Berger MS, McDermott MW, Parsa AT, Vandenberg S, James CD, Lamborn KR, Stokoe D, Haas-Kogan DA. Phase II study of erlotinib plus temozolomide during and after radiation therapy in patients with newly diagnosed glioblastoma multiforme or gliosarcoma. J Clin Oncol. 2009 Feb 1;27(4):579-84. doi: 10.1200/JCO.2008.18.9639. Epub 2008 Dec 15. PMID 19075262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 patients enrolled from 10/2004 - 2/2006. Patients were enrolled at the UCSF Neuro-Oncology clinic.
Groups:
- Temodar Plus Tarceva Plus Radiotherapy: All patients were treated with radiotherapy and temozolomide; patients were treated with dosing of tarceva based upon use of enzyme-inducing antiepileptic drugs
Period: Overall Study
Arm/Group | Temodar Plus Tarceva Plus Radiotherapy
Started | 66
Completed | 65
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Temodar Plus Tarceva Plus Radiotherapy
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Patients were monitored until death
Time Frame: assessment of survival was every 2 months, up to 181 weeks
Population: The analysis was per protocol, and intention to treat. Median overall survival measured from the date of registration was the primary endpoint.
Measure: Median (Full Range); unit: months
Arm/Group | Temodar Plus Tarceva Plus Radiotherapy
Number analyzed (Participants) | 65
months | 19 [3 to 42]

2. Secondary Outcome: Progression Free Survival
Description: Progression based on MR imaging using the Modified McDonnald Criteria defined as 25% increase in sum of products of all measured lesions or any new lesion
Time Frame: every 2 months measure by MR imaging, up to 39 months
Measure: Median (Full Range); unit: months
Arm/Group | Temodar Plus Tarceva Plus Radiotherapy
Number analyzed (Participants) | 65
months | 8.2 [2 to 39]

ADVERSE EVENTS:
Arm/Group | Temodar Plus Tarceva Plus Radiotherapy
Serious Adverse Events (participants affected / at risk) | 2/66
Other Adverse Events (participants affected / at risk) | 4/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temodar Plus Tarceva Plus Radiotherapy (N=66)
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temodar Plus Tarceva Plus Radiotherapy (N=66)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Bone infection NOS (Infections and infestations) | 1 (1)
Cognitive disturbance (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes